CLINICAL TRIAL: NCT05779215
Title: The Multicenter, Prospective, Real-world Registry of Acute Ischemic Stroke With Large- or Medium-vessel Occlusion
Brief Title: Registry of Acute Ischemic Stroke With Large- or Medium-vessel Occlusion
Acronym: LOMEVO
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Junwei Hao, MD, Director of Neurology Department, Xuanwu Hospital, Beijing
Other Study IDs: XMEC-2023-002
Record Dates: First submitted 2023-03-07; First posted 2023-03-22 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; large vessel occlusion; medium vessel occlusion; real-world registry
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute ischemic stroke with large- or medium-vessel occlusion: acute ischemic stroke patients with large- or medium-vessel occlusion including all treatments.
  Interventions: Other: Visit at D90

INTERVENTIONS:
Other: Visit at D90 — Visits at 90±7 days after stroke onset were conducted by trained and blinded investigators, with face-to-face, telephone call or Internet access.

SUMMARY:
This study is designed to observe the treatment options in real-world clinical practice as well as the safety and efficacy of different treatment strategies.

DETAILED DESCRIPTION:
LOMEVO is a prospective, multicenter, real-world registry lasting for 10 years. A total of 50000 patients with large- or medium-vessel occlusion will be enrolled at approximately 30 centers around China.

ELIGIBILITY:
Inclusion Criteria:

* The clinical diagnosis is acute ischemic stroke with large- or medium- vessel occlusion (the criteria followed the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018)
* Informed consent from the patient or surrogate

Exclusion Criteria:

* No additional exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute ischemic stroke due to large- or medium-vessel occlusion will be enrolled and no additional exclusion criteria are set.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2032-04-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) score | 90±7 days
  Ordinal distribution of mRS at 90±7 days; modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)

SECONDARY OUTCOMES:
Excellent functional outcome | 90±7 days
  Proportion of subjects with mRS 0-1 at 90±7 days.
Good functional outcome | 90±7 days
  Proportion of subjects with mRS 0-2 at 90±7 days.
mRS 0-3 | 90±7 days
  Proportion of subjects with mRS 0-3 at 90±7 days.
Change of National Institutes of Health Stroke Scale (NIHSS) | 24 hours
  Change of National Institutes of Health Stroke Scale (NIHSS, a scale between 0 and 42 on which higher scores indicate more severe neurologic deficits) from baseline to 24 hours.
Change of National Institutes of Health Stroke Scale (NIHSS) | 7 days
  Change of National Institutes of Health Stroke Scale (NIHSS, a scale between 0 and 42 on which higher scores indicate more severe neurologic deficits) from baseline to 7 days.
Symptom-to-thrombolysis time (STT) | 24 hours
  Time from onset of symptoms to thrombolytic therapy.
Door-to-Needle Time (DNT) | 24 hours
  Time from the arrival of stroke patient in emergency to initiation of thrombolysis therapy.
Door-to-Puncture Time (DPT) | 24 hours
  Time from the arrival of stroke patient in emergency to groin puncture.
Onset-to-recanalization time | 24 hours
  Time from symptom onset to the beginning of recanalization (recanalization defined as expanded TICI scale≥2b).
Door-to-Recanalization Time (DRT) | 24 hours
  Time from the arrival of stroke patient in emergency to the beginning of recanalization (recanalization defined as expanded TICI scale≥2b).
Puncture-to-recanalization time | 24 hours
  Time from groin puncture to recanalization (recanalization defined as expanded TICI scale≥2b).

OTHER OUTCOMES:
Incidence of clinically significant intracranial hemorrhage | 36 hours
  Incidence of sICH (Heidelberg criteria) measured at 36 hours
Incidence of any intracranial hemorrhage | 36 hours
  Incidence of any intracranial hemorrhage (Heidelberg criteria) measured at 36 hours
All-cause mortality | 90±7 days
  All-cause mortality at 90±7 days
Complications related to intravenous thrombolysis | up to 7 days
  Complications related to intravenous thrombolysis during hospitalization
Complications related to endovascular treatment | up to 7 days
  Complications related to intravenous thrombolysis during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No